CLINICAL TRIAL: NCT04425148
Title: Non-invasive Brain Stimulation for Gamma-induction and Cognitive Enhancement in FTD (Gamma-Induction in FrontoTemporal Dementia, GIFTeD)
Brief Title: Gamma-Induction in FrontoTemporal Dementia Trial
Acronym: GIFTeD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Principal Investigator, Emiliano Santarnecchi, Associate Professor of Radiology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P003553
Record Dates: First submitted 2020-06-01; First posted 2020-06-11 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-02

CONDITIONS: Frontotemporal Dementia
Keywords: FTD
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- tACS (Experimental): 40 Hz transcranial alternating current stimulation (tACS), 30 daily (Monday-Friday) 1-hour sessions
  Interventions: Device: Transcranial Alternating Current Stimulation (tACS)
- Sham tACS (Sham Comparator): Sham transcranial alternating current stimulation (tACS), 30 daily (Monday-Friday) 1-hour sessions
  Interventions: Device: Sham Transcranial Alternating Current Stimulation (sham tACS)

INTERVENTIONS:
Device: Transcranial Alternating Current Stimulation (tACS) — tACS is a noninvasive way of stimulating the brain externally using weak electric currents. Electrodes are placed into a cap that you wear on your head. A weak electrical current travels back and forth through the electrodes to your head.
  Other Names: Non-invasive Brain Stimulation; Neuroelectrics Starstim
  Arms: tACS
Device: Sham Transcranial Alternating Current Stimulation (sham tACS) — Sham (placebo) simulation of transcranial alternating current stimulation without receiving any real stimulation.
  Arms: Sham tACS

SUMMARY:
This is an interventional, sham controlled, double-blind study designed to investigate the safety, tolerability and efficacy of 40 Hz transcranial alternating current stimulation (tACS), a form of noninvasive brain stimulation, delivered for 6 weeks once daily in frontotemporal dementia (FTD) patients. Cognition, gamma EEG activity and brain metabolism via FDG-PET will be measured before and after the tACS intervention.

DETAILED DESCRIPTION:
This is an interventional, multi-site, randomized, double-blind, placebo-controlled study of tACS in patients with FTD. The main aim of this study is to investigate the safety, tolerability and efficacy of gamma-tACS in patients with behavioral variant (bv)-FTD and semantic variant Primary Progressive Aphasia (svPPA), demonstrating tACS potential mechanisms of action, target engagement, and thus informing the design of larger clinical trials.

Participants will be screened at trial sites for determination of eligibility to enter the study on the basis of diagnostic evaluations, according to current diagnostic criteria for probable bv-FTD and safety assessments.

Baseline assessments will consist of behavioral/cognitive evaluations, blood biomarkers, actigraphy, voice biomarkers, EEG and TMS-EEG and tACS with EEG measures, MRI, FDG-PET imaging (5-8 visits). Once participants have met all inclusion and exclusion criteria, they will be randomly assigned to either 6 weeks of daily tACS sessions or 6 weeks of daily Sham tACS sessions.

Post-intervention visits will include FDG-PET scans, MRI, cognitive testing, tACS with EEG, blood biomarkers and TMS-EEG (5-8 visits). A follow-up visit will occur 3 months after the post-invention visit. This visit will include an EEG registration, cognitive testing and behavioral markers.

* tACS is a way of stimulating the brain externally using weak electric currents.

  * Electrodes are placed into a cap that you wear on your head.
  * A weak electrical current travels back and forth through the electrodes to your head.
* FDG-PET is a way of taking pictures of your brain using a special dye that is absorbed into your body. In this study, the dye will help us to see the glucose uptake in your brain. The PET scans for this study will be done at Massachusetts General Hospital (MGH).
* TMS is a noninvasive way of stimulating the brain and will be used in this study to measure your brain's plasticity. Brain plasticity is the brain's ability to change and learn through experience. TMS uses a magnetic field to cause changes in the brain activity. The magnetic field is produced by a coil that is held next to your scalp. We will measure how your brain responds to the TMS before and after the tACS treatment.
* EEG is used in routine clinical care to measure the brain's electrical activity. EEG involves placing a cap with electrodes onto your head.

The investigators will enroll a sample of 20 age-matched healthy controls, who will undergo evaluations similar to the bv-FTD baseline assessment except for PET imaging. Healthy subjects will not have the tACS intervention.

ELIGIBILITY:
FTD Participants

Inclusion Criteria:

* Diagnosis of probable Frontotemporal dementia (bvFTD or svPPA)
* Mini Mental State Examination (MMSE) > 18
* FTLD-specific Clinical Dementia Rating (FTLD-CDR) total score of ≤1
* On stable medications related to cognition or behavior for >30 days such as acetylcholinesterase inhibitors, memantine, anti-depressants, antipsychotic agents, other mood stabilizers, benzodiazepines;
* Age from 40 to 85 years;
* Minimum of completed 8th grade education
* No history of intellectual disability

Exclusion Criteria:

* Current or past history of any significant neurodegenerative disorder of the central nervous system other than FTD e.g. Alzheimer's disease, Lewy body dementia, Parkinson's disease, multiple sclerosis, progressive supranuclear palsy, normal pressure hydrocephalus, Huntington's disease, any condition directly or indirectly caused by Transmissible Spongiform Encephalopathy (TSE), Creutzfeldt-Jakob Disease (CJD), variant Creutzfeldt-Jakob Disease (vCJD), or new variant Creutzfeldt-Jakob Disease (nvCJD);
* Current or past history of stroke (cortical stroke), intracranial brain lesions, previous neurosurgery or head trauma that resulted in residual neurologic impairment.

  * Non-cortical disease such as confluence white matter changes (including lacunar infarcts < 1cm) and asymptomatic, subacute, cerebellar infarcts may be included upon review of a medically responsible neurologist.
* Past or current history of major depression, bipolar disorder, psychotic disorders, or any other major psychiatric condition will be evaluated by the study MD.
* Current history of poorly controlled migraines including chronic medication for migraine prevention
* History of seizures with the exception of a single seizure of benign etiology (e.g. febrile seizure) in the judgment of the investigator;
* History of fainting spells of unknown or undetermined etiology that might constitute seizures.
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.).
* Metal implants in the head (except dental), pacemaker, medication pump, nerve stimulator, TENS unit, ventriculo-peritoneal shunt, cochlear implant, unless cleared by the study MD.
* Contraindication for undergoing MRI or receiving TMS or tACS;
* Any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included;
* >50 mSv of radiation exposure for research within the past year (PET imaging exclusion);
* Substance abuse or dependence within the past six months;
* Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following: The patient's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination of CNS active drugs;
* All female participants that are pre-menopausal will be required to have a pregnancy test; any participant who is pregnant or breastfeeding will not be enrolled in the study;
* Subjects who, in the investigator's opinion, might not be suitable for the study;
* A hair style or head dress that prevents electrode contact with the scalp or would interfere with the stimulation (for example: thick braids, hair weave, afro, wig).

Healthy Volunteers

Inclusion Criteria:

* Age: 40-85 years
* Normal healthy volunteer
* Right-handed (assessed by means of the Edinburgh Handedness Questionnaire)
* MMSE >27
* Minimum of completed 8th grade education
* No history of intellectual disability

Exclusion Criteria:

* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG or family history of treatment resistant epilepsy, with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of the investigator
* History of head injury resulting in prolonged loss of consciousness
* Any metal in the brain, skull or elsewhere unless approved by the responsible MD
* Any medical devices (i.e. Cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible MD
* Past or current history of major depression, bipolar disorder or psychotic disorders, or any other major psychiatric condition.
* Neurological disorder or intracranial lesion (including an incidental finding on MRI)
* Current history of poorly controlled migraines including chronic medication for migraine prevention
* Any unstable medical condition
* Pregnancy
* Medications will be reviewed by the responsible MD and a decision about inclusion will be made based on the following:

  * The participant's past medical history, drug dose, history of recent medication changes or duration of treatment, and combination with other CNS active drugs.
* Substance abuse or dependence within the past six months
* Subjects who, in the investigator's opinion, might not be suitable for the study
* Diseased or damaged skin over the face or scalp
* A hair style or head dress that prevents electrode contact with the scalp (for example: thick braids, hair weave, afro, wig)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Attrition (withdrawal) rate | up to 6 months
  The rate of enrolled participants who withdraw from the study will be reported
Change in Gamma activity | up to 6 months
  Changes in oscillatory activity in the EEG gamma band will be evaluated before and after the tACS sessions
Change in Cognition | up to 6 months
  Change in Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) score will be reported. The score ranges from 0-85 with the higher score meaning greater cognitive impairment.
Change in Cognition | up to 6 months
  Change in Frontal Assessment Battery (FAB) score will be reported. The scores range from 0-18 with a higher score meaning less cognitive impairment.
Change in Brain Metabolism measured via FDG-PET | up to 3 months
  Change in brain glucose metabolism will be measured via FDG-PET after the daily tACS sessions

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Santarnecchi, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States
- Fondazione Santa Lucia, Roma, Italy

IPD SHARING:
Plan to Share IPD: No